CLINICAL TRIAL: NCT00860899
Title: Postoperative Pain and Systemic Inflammatory Stress Response (SIRS) After Preoperative Analgesia With Clonidine or Levobupivacaine
Brief Title: Postoperative Pain and SIRS After Preoperative Analgesia With Clonidine or Levobupivacaine
Acronym: PPSAPACL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital Dubrava (Other)
Responsible Party: Principal Investigator, Jasminka Persec, MD, PhD, MD PhD, University Hospital Dubrava
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1860; 1861
Record Dates: First submitted 2009-03-10; First posted 2009-03-12 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Analgesia; Pain; Systemic Inflammatory Stress Response
Keywords: clonidine; levobupivacaine; preoperative analgesia; postoperative pain; systemic inflammatory stress response; epidural analgesia; Anesthetics, Local
MeSH Terms: conditions — Agnosia; Pain; Pain, Postoperative | interventions — Clonidine; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- clonidine (Active Comparator): Clonidine is an alpha2-adrenergic agonist with sedative, analgesic and hemodynamic properties. It inhibits transmission of nociceptive stimuli in the dorsal horn of the spinal cord, acting on the inhibitory descending pathways.
  Interventions: Drug: clonidine, levobupivacaine
- levobupivacaine (Active Comparator): Levobupivacaine is long-acting local anesthetic, S-enantiomer of bupivacaine, with identical anesthetic potency.
  Interventions: Drug: clonidine, levobupivacaine

INTERVENTIONS:
Drug: clonidine, levobupivacaine — One hour prior to skin incision, on epidural catheter, patients received 5 µg/kg of clonidine [Catapres®, Boehringer Ingelheim, Germany], 7 mL of 0.25% levobupivacaine [Chirocaine®, Abbott S.p.A., Italy] or 7 mL of saline.The study was designed to compare clonidine and levobupivacaine, and than both with the control group, in order to asses their analgesic and immunomodulation efficacy.
  Other Names: clonidine [Catapres®, Boehringer Ingelheim, Germany]; levobupivacaine [Chirocaine®, Abbott S.p.A., Italy]

SUMMARY:
The purpose of this study was to investigate hypothesis that preoperative administration of epidural clonidine will reduce postoperative pain and systemic inflammatory stress response better than epidural levobupivacaine.

DETAILED DESCRIPTION:
Investigations showed that upregulation of prostaglandin E2 and interleukin-6 at central sites is an important component of surgery induced inflammatory response in patients. Postoperative period is associated with an increased production of cytokines, which augment pain sensitivity. With adequate perioperative pain control it is possible to control central and peripheral inflammatory response to surgery, and influence on patient outcomes. Use of analgetics before the pain stimulus (preventive analgesia) prevent development of neuroplastic changes in central nervous system, and reduces pain. Clonidine is an alpha2-adrenergic agonist with sedative, analgesic and hemodynamic properties. It inhibits transmission of nociceptive stimuli in the dorsal horn of the spinal cord, acting on the inhibitory descending pathways. According to recent experimental investigations clonidine lowers proinflammatory cytokine level, and prevents hypersensitization acting through adrenoreceptors alpha-2A.

Levobupivacaine is a long-acting local anesthetic, S-enantiomer of bupivacaine, with identical anesthetic potency. When administered intraperitoneally or by local infiltration of operation site, levobupivacaine produced analgesia and reduction of proinflammatory cytokines. Investigations of epidural and intrathecal levobupivacaine provide evidence for improved postoperative analgesia with reduced analgesic consumption. But, it remains unknown if that analgesia is sufficient enough to blockade inflammatory stress response during perioperative time.We want to investigate and compare analgesic and immunomodulation efficacy of this two frequently used analgesics.

ELIGIBILITY:
Inclusion Criteria:

* colorectal resection surgery patients
* preoperative risk of anesthesia and operation, ASA (American Society of Anesthesiologists) physical status I or II

Exclusion Criteria:

* diabetes mellitus
* renal insufficiency
* liver insufficiency
* autoimmune disease
* corticosteroid and immunosuppressive use
* operation time exceeding six hours

Ages: 42 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
postoperative pain level | 1 h before surgery, 1 h after start of the surgery, 1 h , 6 h , 12 h and 24 h after surgery

SECONDARY OUTCOMES:
systemic inflammatory stress response | 1 hour before surgery, 1 hour after start of the surgery, 1 h , 6 h , 12 h and 24 h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jasminka Persec, MD PhD, Principal Investigator — Anesthesiology, Resuscitation and Intensive Care Medicine Clinic, University Hospital Dubrava; Zoran Persec, MD Msc, Study Chair — Department of Urology, University Hospital Dubrava; Ino Husedzinovic, Prof. MD PhD, Study Director — Anesthesiology, Resuscitation and Intensive Care Medicine Clinic, University Hospital Dubrava
Locations (1):
- University Hospital Dubrava, Zagreb, Croatia

REFERENCES:
- [Background] 1. Buvanendran A, Kroin JS, Berger RA, Hallab NJ, Saha C et al.Anesthesiology 104(3):403-410, 2006. 2. Katz J. Curr Opin Anaesthesiol 15(4):435-441, 2002. 3. Carr DB. Anesthesiology 85(6): 1498-1499, 1996. 4. Lavand'homme PM, Eisenach JC. Pain 105(1-2):247-254, 2003. 5. Nader ND, Ignatowski TA, Kurek CJ, Knight PR, Spengler RN. Anesth Analg 93(2):363-369, 2001. 6. Wu CT, Jao SW, Borel CO, Yeh CC, Li CY, Lu CH et al. Anesth Analg 99(2):502-509, 2004. 7. Novak-Jankovic V, Bovill JG, Ihan A, Osredkar J. Eur J Anaesthesiology 17(1):50-56, 2000. 8. Kim MH, Hahn TH. Anesth Analg 90(6):1441-1444, 2000. 9. Louizos AA, Hadzilia SJ, Leandros E, Kouroukli IK, Georgiou LG et al. Surg Endosc 19(11):1503-1506, 2005. 10. Meisner M, Brunkhorst FM, Reith HB, Schmidt J, Lestin HG et al. Clin Chem Lab Med 38(10):989-995, 2000. 11. Naeini AE, Montazerolghaem S. Saudi Med J 27(3):422-424, 2006. 12. Sarbinowski R, Arvidsson S, Tylman M, Oresland T, Bengtsson A. Acta Anaesthesiol Scand 49(2):191-196, 2005.